CLINICAL TRIAL: NCT01204541
Title: A Single-Center Pilot Study to Assess Macular Function
Status: Completed | Type: Observational
Sponsor: ORA, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 10-120-0013
Record Dates: First submitted 2010-09-16; First posted 2010-09-17 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Macular Degeneration
Keywords: Non-exudative age-related macular degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- AMD
- Young normals
- Older normals

SUMMARY:
This study seeks to evaluate a novel endpoint for future dry AMD clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Subjects in good health aged 20-29 or 60-90 years (normal cohorts)
* Subjects with early non-exudative age-related macular degeneration (AMD cohort)

Exclusion Criteria:

* Enrollment in a investigational drug or device study and have used an investigational drug or device within 7 days of enrollment into this study

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Three groups of subjects will be enrolled:
  1. Normal healthy subjects aged 20-29 years
  2. Normal healthy subjects aged 60-90 years
  3. Subjects with early dry AMD
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2010-09; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Andover, Massachusetts, United States